CLINICAL TRIAL: NCT00486837
Title: Multicenter, Randomized, Parallel Group Study to Investigate the Optimal Deposition Site for Inhaled Prolastin® in Patients With Cystic Fibrosis (CF)
Brief Title: Deposition of Inhaled Prolastin in Cystic Fibrosis Patients
Acronym: CF2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100452
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Bronchial Deposition Intervention: Alpha1-Proteinase Inhibitor (Human) Dosage: 25 mg in lungs, one inhalation per day over 4 weeks
  Interventions: Drug: Alpha1-Proteinase Inhibitor (Human)
- Group 2 (Experimental): Peripheral Deposition Intervention: Alpha1-Proteinase Inhibitor (Human) Dosage: 25 mg in lungs, one inhalation per day over 4 weeks
  Interventions: Drug: Alpha1-Proteinase Inhibitor (Human)

INTERVENTIONS:
Drug: Alpha1-Proteinase Inhibitor (Human) — 25 mg of Alpha1-Proteinase Inhibitor (Human) in the lungs, one inhalation per day over 4 weeks.
  Other Names: Prolastin®; Alpha-1 antitrypsin (AAT); BAY x 5747; BAY 10-5233; TAL-05-00007; A1AT; NDC 13533-601-30; NDC 13533-601-35

SUMMARY:
The objective of this trial is to determine the optimal region of the lung for depositing Prolastin (alpha-1 antitrypsin; AAT) by inhalation in order to treat cystic fibrosis (CF). The AKITA® nebulizer has settings which can be varied to target the inhaled drug to either the deep lung or to the upper airways in a one to one randomization. The study will measure how much of the activity of the enzyme elastase is inhibited by AAT.

DETAILED DESCRIPTION:
The optimum deposition site (bronchial or peripheral) in CF patients for AAT will be investigated by measuring several parameters in induced sputum. The study will start with a 2 week run-in period in which the planned 60 patients inhale isotonic saline once daily. This period is followed by a 4 week treatment period where 30 patients inhale AAT for peripheral deposition and 30 patients inhale AAT for bronchial deposition. Six patients in each group will be asked to collect spontaneous sputum at home.

Twenty-five milligrams of AAT will be deposited at one of the two target sites using the AKITA® device. The inhalation should take place in the evening between 18.00 and 23.00 h.

Patients will inhale saline once daily for 2 weeks (run-in period) followed by 4 weeks of once daily inhalation of AAT. Induced sputum will be collected at visits to the clinic at the start of the run-in, at the start of AAT treatment, and at 2 and 4 weeks after the start of AAT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of CF
* Age >= 8 years
* Forced expiratory volume at one second (FEV1) > 25 % of predicted value
* Free elastase activity checked at visit 1 must be positive (free elastolytic activity in the sample, 2 standard deviations above of the negative blank samples in the assay.) .
* Patient must be positive at least 3 times for pseudomonas in the last 2 years
* Patient must be positive for pseudomonas at Visit 1
* Patient must be able to perform reliable spirometry
* Patient must be on stable concomitant therapy at least 2 weeks prior to visit 1 and during the study
* Written informed consent of the patient or legal representative(s)

Exclusion Criteria:

* FEV1 < 25% of predicted value post-bronchodilator
* History of lung transplant
* Any lung surgery within the past 2 years
* On any thoracic surgery waiting list
* Severe concomitant disease (serious malignant disease, congestive heart failure New York Heart Association (NYHA) III/IV, cor pulmonale with the need of oxygen therapy)
* Severe liver cirrhosis with ascites, hypersplenism or grade III/IV esophageal varices.
* Known selective immunoglobulin A (IgA) deficiency with known antibody against IgA (anti-IgA antibody)
* Active pulmonary exacerbation within the 4 weeks prior to screening
* Current Smoking
* Pregnancy or lactation
* Women of child-bearing age without adequate contraception
* Any medical condition which the investigator feels will prohibit the patient from completing the trial
* Participation in another clinical trial within 30 days prior to inclusion at visit 1

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-12; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Griese, MD, Principal Investigator — Kinderklinik und Kinderpoliklinik im Haunerschen Kinderspital

REFERENCES:
- [Result] Griese M, Latzin P, Kappler M, Weckerle K, Heinzlmaier T, Bernhardt T, Hartl D. alpha1-Antitrypsin inhalation reduces airway inflammation in cystic fibrosis patients. Eur Respir J. 2007 Feb;29(2):240-50. doi: 10.1183/09031936.00047306. Epub 2006 Oct 18. PMID 17050563
- See also: FDA Approved Product Labeling Information — http://www.talecris-pi.info/inserts/Prolastin.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed in 8 study centers in Germany.
Pre-assignment Details: Subjects inhaled saline once daily for 2 weeks during the Run-in Period.
Groups:
- Peripheral Deposition: Peripheral Deposition is achieved with a breathing maneuver consisting of slow and deep breaths
- Bronchial Deposition: Bronchial Deposition consists of inhalation of smaller volumes per breath at higher flow rates
Period: Overall Study
Arm/Group | Peripheral Deposition | Bronchial Deposition
Started | 37 | 35
Completed | 28 | 28
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — No sputum, devise issues, exacerbation | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Deposition | Bronchial Deposition | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.78 (7.54) | 27.42 (9.78) | 25.46 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Germany | 37 | 35 | 72
Free Elastase during the Run-In Phase [Mean (Standard Deviation); unit: µg/mL]
  Week 0 | 36.6 (35.9) | 35.9 (38.8) | 36.2 (36.9)
  Week 2 | 32.7 (31.7) | 25.0 (20.1) | 29.1 (27.0)
  Absolute Change | -4.0 (21.3) | -10.9 (36.9) | -7.25 (29.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Free Elastase in Induced Sputum From Baseline to Week 4
Time Frame: Baseline vs Week 4
Population: Modified Intent-to-Treat Population (mITT) was all randomized subjects who received any amount of study medication and had at least one evaluation of the primary efficacy variable (free elastase in induced sputum) post baseline and at baseline (Visit 2).
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Peripheral Deposition | Bronchial Deposition
Number analyzed (Participants) | 28 | 24
ug/mL | -7.42 (29.96) | 6.11 (31.30)
Statistical Analysis 1: Comparison: Peripheral Deposition vs Bronchial Deposition; Test type: Superiority or Other; p = 0.197, ANCOVA

2. Secondary Outcome: Change in Alpha-1-anti-trypsin (A1AT) Activity in Induced Sputum From Baseline at Week 4
Time Frame: Baseline vs Week 4
Population: For Group 1, only 24 out of 28 subjects had applicable data to analyze. For Group 2, only 27 out of 28 subjects had applicable data to analyze.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Group 1: Bronchial Deposition
  Alpha1-Proteinase Inhibitor (Human): 25 mg of Alpha1-Proteinase Inhibitor (Human) in the lungs, one inhalation per day over 4 weeks.
- Group 2: Peripheral Deposition
  Alpha1-Proteinase Inhibitor (Human): 25 mg of Alpha1-Proteinase Inhibitor (Human) in the lungs, one inhalation per day over 4 weeks.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 27
ug/mL | 16741 (33583) | 6469 (18999)

3. Secondary Outcome: Change in Total Immunoglobulin G (IgG) Fragments in Induced Sputum From Baseline at Week 4
Time Frame: Baseline vs Week 4
Population: For Group 1, only 24 out of 28 subjects had applicable data to analyze. For Group 2, only 26 out of 28 subjects had applicable data to analyze.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 26
ug/mL | 0.005 (1.10) | -0.48 (1.53)

4. Secondary Outcome: Change in Total Bacterial Load in Induced Sputum From Baseline to Week 4
Time Frame: Week 4
Population: For Group 1, only 24 out of 28 subjects had applicable data to analyze. For Group 2, all 28 subjects had applicable data to analyze.
Measure: Mean (Standard Deviation); unit: CFU/g
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 28
CFU/g | 22673275.8 (253455845.23) | 5021353.2 (130686274.77)

5. Secondary Outcome: Change in Pseudomonas Load in Induced Sputum From Baseline at Week 4
Time Frame: Baseline vs Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: CFU/g
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 24 | 28
CFU/g | -40.1 (808.2) | -22.3 (772.4)

6. Secondary Outcome: Change in Neutrophil Number in Induced Sputum From Baseline at Week 4
Time Frame: Baseline vs Week 4
Population: For Group 1, only 21 out of 28 subjects had applicable data to analyze. For Group 2, only 22 out of 28 subjects had applicable data to analyze.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 21 | 22
percentage of change | -20.8 (30.3) | -8.2 (20.9)

ADVERSE EVENTS:
Arm/Group | Peripheral Deposition | Bronchial Deposition
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 10/37 | 13/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peripheral Deposition (N=37) | Bronchial Deposition (N=35)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 5
Sinusitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the Investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.